CLINICAL TRIAL: NCT04910269
Title: An International Multicenter, Randomized, Double-Blind, Placebo-Controlled Trial of the Safety and Efficacy of Anti-Coronavirus Hyperimmune Intravenous Immunoglobulin for the Treatment of Adult Outpatients in Early Stages of COVID-19
Brief Title: Outpatient Treatment With Anti-Coronavirus Immunoglobulin
Acronym: OTAC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institutes of Health (NIH) (NIH); International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INSIGHT12; 2021-001663-24 (EudraCT Number)
Record Dates: First submitted 2021-06-01; First posted 2021-06-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: COVID; SARS-CoV2 Infection; Covid19
Keywords: immunotherapy; hIVIG; early treatment
MeSH Terms: conditions — COVID-19 | interventions — HIV hyperimmune globulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants in this group will receive the investigational treatment in addition to standard of care.
  Interventions: Biological: Hyperimmune immunoglobulin to SARS-CoV-2 (hIVIG)
- Placebo Group (Placebo Comparator): Participants in this group will receive a placebo in addition to standard of care.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Hyperimmune immunoglobulin to SARS-CoV-2 (hIVIG) — The hIVIG product is administered as a single dose of 3.5 grams, or 35 milliliter at a concentration of 0.1 grams/milliliter.
  Arms: Treatment Group
Other: Placebo — Infusion of 35 milliliters standard isotonic saline
  Arms: Placebo Group

SUMMARY:
The primary objective of the Outpatient Treatment with Anti-Coronavirus Immunoglobulin (OTAC) (INSIGHT 012) trial is to compare the safety and efficacy of a single infusion of anti-COVID-19 hyperimmune intravenous immunoglobulin (hIVIG) versus placebo among adults with recently diagnosed severe acute respiratory syndrome - coronavirus 2 (SARS-CoV2) infection who do not require hospitalization. The primary endpoint of this double-blind randomized trial is a five-category ordinal outcome that assesses the participant's clinical status seven days after the infusion of hIVIG or placebo.

1. Asymptomatic and no limitations in usual activity due to COVID-19
2. Mild COVID-19 illness or minor limitations to usual activity
3. Moderate COVID-19 illness and with major limitations to usual activity
4. Severe COVID-19 or serious disease manifestation from COVID-19
5. Critical illness from COVID-19 or Death

Two strata of participants will be identified for analysis purposes. Stratum 2 will be participants who receive direct-acting antivirals (DAAs) or other anti-SARS-CoV2 agents that are approved/available and recommended for use as part of standard of care (SOC), estimated to be about 20% of participants. Stratum 1 will be participants who do not receive this agents, estimated to be about 80% of participants.

DETAILED DESCRIPTION:
The primary objective will be addressed by testing two hypotheses aimed at assessing whether hIVIG + standard of care (SOC) is superior to placebo + SOC for the primary ordinal endpoint at Day 7. These hypotheses will be tested for the following two groups: a) among all randomized participants (stratum 1 and 2), and b) among only participants enrolled in stratum 1. For the primary analysis, overall type 1 error will be controlled at 5% by using a 2-sided significance level of 0.035 for each hypothesis. This significance level was obtained using the correlation between the test statistics for the proportional log odds ratio for all randomized participants and for this log odds ratio for those in stratum 1. This correlation was determined to be 0.895. With this approach hIVIG will be considered superior to placebo if either of the two hypotheses is rejected.

Participants will be randomized to a single infusion of an hIVIG product or placebo in a 1:1 allocation. Randomization will be stratified by study site pharmacy and the two SOC strata.

ELIGIBILITY:
Inclusion Criteria:

* Clinical risk based on age ≥ 55 years or an adult (age ≥ 18 years) with an immunosuppressed condition.
* Positive test for SARS-CoV-2 within ≤5 days (if >1 test, the first positive is within ≤5 days). Tests may include an institutional-based nucleic acid amplification test (NAAT), or any protocol-approved rapid test.
* Within ≤5 days from symptom onset, if symptomatic from current SARS-CoV-2 infection.
* Agrees to not participate in another clinical trial for the treatment or management of SARS-CoV-2 infection through Day 7, or until hospitalized or significant disease progression if prior to Day 7 (defined by ordinal category 4 or 5).
* Participant provides written informed consent prior to study procedures, and understands and agrees to adhere to planned study procedures through Day 28.

Ongoing immunosuppressive condition or immunosuppressive treatment, includes:

1. Steroids equivalent to prednisone > 10 mg/day for at least the last 28 days
2. Rheumatologic or autoimmune disorder treated with a biologic or non-biologic immunosuppressive therapy
3. Antirejection medicine after solid organ or stem cell transplantation
4. Cancer treatment with systemic chemotherapy, biologic and/or cell-based therapy in the last 12 months
5. Primary or acquired severe B- or T-lymphocyte immune dysfunction
6. HIV infection
7. Splenectomy or functional asplenia

Exclusion Criteria:

* Asymptomatic and had prior symptoms from the current infection that have now resolved (for >24 hours).
* Asymptomatic and has received a vaccination for COVID-19 (≥1 dose).
* Undergoing evaluation for possible admission to hospital for medical management (this does not include evaluation of possible hospitalization for public health purposes).
* Evidence of pneumonia and/or hypoxia due to COVID-19 (NOTE: chest imaging is not required, but if available it should not show new infiltrates suggestive of pneumonia; hypoxia is defined by new oxygen supplementation or increase above pre-illness level).
* Prior receipt of immunoglobulin product or passive immune therapy for SARS-CoV-2 in the past 90 days (i.e., convalescent plasma, SARS-CoV-2 monoclonal antibodies, or any IVIG).
* Any of the following thrombotic or procoagulant conditions or disorders:

  1. acute coronary syndrome, cerebrovascular syndrome, pulmonary embolism, or deep venous thrombosis within 28 days of randomization.
  2. prothrombin gene mutation 20210, homozygous Factor V Leiden mutations, antiphospholipid syndrome, or a deficiency in antithrombin III, protein C, or protein S.
* History of hypersensitivity to blood, plasma or IVIG excipients.
* Known immunoglobulin A (IgA) deficiency or anti-IgA antibodies.
* In the opinion of the investigator, any condition for which participation would not be in the best interest of the participant or that could prevent or confound protocol assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Status | 7 days
  The primary outcome is to compare the safety and efficacy of a single infusion of hIVIG versus placebo on clinical status after seven days. Outcome will be reported as the percent of participants who fall into each of 5 clinical status categories as defined below.
  1. Asymptomatic and no limitations in usual activity due to COVID-19
  2. Mild COVID-19 illness or minor limitations to usual activity
  3. Moderate COVID-19 illness and with major limitations to usual activity
  4. Severe COVID-19 or serious disease manifestation from COVID-19
  5. Critical illness from COVID-19 or Death

SECONDARY OUTCOMES:
All-cause hospitalization or death through 28 days. | 28 days
  Outcome reported as the percent of participants who are hospitalized or who expire for any reason by day 28 post treatment.
All-cause mortality through 28 days. | 28 days
  Outcome reported as the percent of participants who expire for any reason by day 28 post treatment.
Significant Disease Progression | 28 days
  Outcome is reported as the number of participants with significant disease progression through 28 days, which is defined by fulfilling criteria for category 4 or 5 on the ordinal scale using a time to event analysis.
Ordinal Scale Distribution | 4, 14, 28 days
  Outcome will be reported as the percent of participants who fall into each of 5 clinical status categories as defined below at days 4, 14, and 28 following treatment.
  1. Asymptomatic and no limitations in usual activity due to COVID-19
  2. Mild COVID-19 illness or minor limitations to usual activity
  3. Moderate COVID-19 illness and with major limitations to usual activity
  4. Severe COVID-19 or serious disease manifestation from COVID-19
  5. Critical illness from COVID-19 or Death
Disease Progression Through 7 Days | 7 days
  Outcome is reported as the proportion of participants with any disease progression at Day 7, using a sliding dichotomous scale progression defined by a categorization on the ordinal scale that is worse than the status at entry.
Significant Disease Progression Through 7 Days | 7 days
  Outcome is reported as the proportion of participants who progress to categories 3-5 on the clinical ordinal scale at Day 7 among participants in categories 1 or 2 of the ordinal scale at entry.
Disease Progression at Follow-up | 7, 14, 28 days
  Outcome is reported as the percent of participants who experience severe disease progression during follow-up, defined by the worst health status achieved on the clinical ordinal scale at any point by Day 7, 14, and 28.
Activity Limitations at Follow-up | 7, 14, 28 days
  Outcome is reported as the percent of participants who attain their pre-COVID health status without limitations in usual activity (defined as category 1 on the ordinal scale) at Day 7, 14, and 28.
Change in Viral Burden from Serum Antigen | 7 days
  Outcome is reported as the change between Day 0 and Day 7 in viral burden as determined by serum antigen levels from nasal and saliva specimens.
Change in Viral Burden from PCR | 7 days
  Outcome is reported as the change between Day 0 and Day 7 in viral burden as determined by polymerase chain reaction (PCR) from nasal and saliva specimens.
Change in SARS-CoV-2 Antibody Concentration | 7 days
  Outcome is reported as the change in SARS-CoV-2 antibody levels between Day 0 and Day 7, including subclasses and neutralizing titers.
Healthcare Utilization at Follow-up | 28 days
  Outcome is reported as the percent of participants who had health care engagement for the purposes of medical evaluation and/or management of COVID-19 illness (e.g., via telehealth, clinic, urgent care, emergency room, or hospitalization) at 28 days follow-up.
Worst Status Through 28 Days | 28 days
  Outcome is reported as the number of participants who experience each of the following categories as their worst respiratory status through 28 days, including: a) no respiratory symptoms, b) upper respiratory symptoms, c) lower respiratory symptoms without hypoxia, c) hypoxia requiring conventional oxygen supplementation by nasal canula, d) respiratory failure requiring high-flow oxygen delivery device or non-invasive ventilation, or e) respiratory failure requiring mechanical ventilation or extra-corporeal membrane oxygenation (ECMO).
Hypoxemia Through Day 7 | 7 days
  Outcome is reported as the mean oxygen saturation (percentage) level in each group at 7 days.
Additional COVID-19 Treatment | 28 days
  Outcome is reported as the number of patients starting other treatments targeting COVID-19 through 28 days post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Cavan Reilly, PhD, Principal Investigator — University of Minnesota
Locations (65):
- United States (22):
  - Southern Arizona VA Healthcare System (074-009), Tucson, Arizona
  - VA Northern California Health Care System (074-023), Mather, California
  - Stanford University Hospital & Clinics (Site 203-003), Palo Alto, California
  - San Francisco VAMC (Site 074-002), San Francisco, California
  - Rocky Mountain Regional VA Medical Center (074-010), Aurora, Colorado
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Washington DC Veterans Affairs Medical Center, Washington D.C., District of Columbia
  - University of Maryland Medical System, Baltimore, Maryland
  - Henry Ford Health System Site (014-001), Detroit, Michigan
  - Infusion Associates, Grand Rapids, Michigan
  - Mount Sinai Beth Israel Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Foundation (Site 207-001), Cleveland, Ohio
  - Penn State Health Milton S. Hershey Medical Center (209-002), Hershey, Pennsylvania
  - Hendrick Medical Center, Abilene, Texas
  - CHRISTUS Spohn Shoreline Hospital, Corpus Christi, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Intermountain Medical Center (211-001), Murray, Utah
  - UVA Health System, University Hospital (Site 210-003), Charlottesville, Virginia
  - Carilion Medical Center (Site 080-018), Roanoke, Virginia
  - Salem VA Medical Center (074-014), Salem, Virginia
  - Swedish Hospital First Hill, Seattle, Washington
- Argentina (4):
  - Instituto Medico Platense, La Plata, Buenos Aires
  - Centro de Investigaciones Medicas de Mar del Plata (Site 611-031), Mar del Plata, Buenos Aires
  - Clínica Central S.A. (611-028), Villa Regina, Río Negro Province
  - Hospital General de Agudos JM Ramos Mejia, Buenos Aires
- St. Vincent's Hospital, Sydney, New South Wales, Australia
- Denmark (8):
  - Odense University Hospital, Odense, C
  - Aarhus Universitetshospital, Skejby, Aarhus, N
  - Department of Infectious Diseases, Aalborg
  - Rigshospitalet, CHIP, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Herlev/Gentofte Hospital, Hellerup
  - Hvidovre University Hospital, Department of Infectious Diseases, Hvidovre
  - Kolding Sygehus, Kolding
- Greece (5):
  - Dept of Critical Care and Pulmonary Medicine, Evangelismos General Hospital, Athens, Attica
  - 3rd Dept of Medicine, Medical School, Athens, Attica
  - Laiko Athens General Hospital, Athens, Attica
  - Department of Clinical Therapeutics of Alexandra Hospital, Athens, Attica
  - 4th Department of Internal Medicine, Athens, Attica
- India (2):
  - All India Institute of Medical Sciences (AIIMS), Jodhpur, Rajasthan
  - Postgraduate Institute of Medical Education and Research (PGIMER), Chandigarh
- Mexico (5):
  - Hospital General Dr. Manuel Gea Gonzáles, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias Ismael Cosió Villegas, Mexico City, Mexico City
  - CHRISTUS Centro de Excelencia en Investigacion (Obispado), Monterrey, Nuevo León
  - Hospital General Dr. Aurelio Valdivieso, Oaxaca City, OA
- Unidad de Ensayos Clinicos Socios En Salud Sucursal Perú (651-009), Lima, Peru
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - CAP Can Bou, Castelldefels, Barcelona
  - CAP El Maresme, Mataró, Barcelona
  - CAP Corbera, Barcelona
- Thailand (4):
  - Siriraj Hospital (Site 613-002), Bangkok Noi, Bangkok
  - Chulalongkorn University and The HIV-NAT, Pathum Wan, Bangkok
  - Khon Kaen University, Srinagarind Hospital (Site 613-003), Khon Kaen
  - Bamrasnaradura Infections Diseases Institute (613-007), Nonthaburi
- Uganda (6):
  - MRC/UVRI & LSHTM Uganda Research Unit, Entebbe
  - Joint Clinical Research Center (JCRC), Kampala
  - Makerere University Lung Institute (Site 634-604), Kampala
  - St. Francis Hospital, Nsambya, Kampala
  - Lira Regional Referral Hospital, Lira
  - Masaka Regional Referral Hospital, Masaka
- Central City Clinical Hospital of Ivano-Frankivsk City Council, Ivano-Frankivsk, Ukraine
- United Kingdom (2):
  - University College London Hospitals, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
A public data set will be made available at the end of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Jha A, Barker D, Lew J, Manoharan V, van Kessel J, Haupt R, Toth D, Frieman M, Falzarano D, Kodihalli S. Efficacy of COVID-HIGIV in animal models of SARS-CoV-2 infection. Sci Rep. 2022 Oct 10;12(1):16956. doi: 10.1038/s41598-022-21223-2. PMID 36216961